CLINICAL TRIAL: NCT01008098
Title: Neuroprotective/Neurotrophic Effect of Lexapro® in Patients With Posttraumatic Stress Disorder
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, In Kyoon Lyoo, MD, PhD, MMS, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KR_12661A
Record Dates: First submitted 2009-11-03; First posted 2009-11-05 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; Escitalopram; Magnetic Resonance Imaging; BDNF
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PTSD group (Experimental)
  Interventions: Drug: escitalopram (lexapro)

INTERVENTIONS:
Drug: escitalopram (lexapro) — 0 - 4 week: 10 mg escitalopram a day 5 - 8 week: 20 mg escitalopram a day

SUMMARY:
The objectives of the current study are

1. to evaluate the efficacy of escitalopram in treatment for post-traumatic stress disorder,
2. to find the structural changes of brain using magnetic resonance imaging and its association with the symptoms reduction, and
3. to look at the differences of brain imaging findings and symptoms changes according to genetic differences of brain-derived neurotrophic factor (a biological molecule facilitating neuronal growth in human).

ELIGIBILITY:
Inclusion Criteria:

* 18-65 year-old male or female
* PTSD diagnosed by SCID-IV

Exclusion Criteria:

* Previous or current treatment history for PTSD
* Neurologic disease (eg., epilepsy, infarct, multiple sclerosis, brain tumor)
* Any other axis I psychiatric disorder diagnosed by SCID-IV
* Borderline personality disorder or antisocial personality disorder
* IQ below 80
* Any contraindication to MRI scan
* Any current psychotropic medication
* Unstable medical illness or severe abnormality in laboratory test at screening assessment
* Women who are pregnant, breastfeeding, or planning pregnancy
* Any contraindications to drug used in the study (e.g., allergy, intolerance, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2008-11; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in brain structure, function, and biochemical metabolism, analyzed using the computational approach | Baseline, 8th weeks
Change from baseline in Clinician-administered PTSD scale scores at 1st week | Baseline, 1st week
Change from baseline in Clinician-administered PTSD scale scores at 4th weeks | Baseline, 4th weeks
Change from baseline in Clinician-administered PTSD scale scores at 8th weeks | Baseline, 8th weeks

SECONDARY OUTCOMES:
Change from baseline in Hamilton depression rating scale scores at 1st week | Baseline, 1st week
Change from baseline in Hamilton anxiety rating scale scores at 1st week | Baseline, 1st week
Number of participants with adverse events | 1st week
Change from baseline in Hamilton depression rating scale scores at 4th weeks | Baseline, 4th weeks
Change from baseline in Hamilton depression rating scale scores at 8th weeks | Baseline, 8th weeks
Change from baseline in Hamilton anxiety rating scale scores at 4th weeks | Baseline, 4th weeks
Change from baseline in Hamilton anxiety rating scale scores at 8th weeks | Baseline, 8th weeks
Number of participants with adverse events | 4th weeks
Number of participants with adverse events | 8th weeks

CONTACTS AND LOCATIONS:
Overall Officials: In Kyoon Lyoo, MD, PhD, MMS, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea